CLINICAL TRIAL: NCT03449446
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of Selonsertib, GS-0976, GS-9674, and Combinations in Subjects With Bridging (F3) Fibrosis or Compensated Cirrhosis (F4) Due to Nonalcoholic Steatohepatitis (NASH)
Brief Title: Study to Evaluate the Safety and Efficacy of Selonsertib, Firsocostat, Cilofexor, and Combinations in Participants With Bridging Fibrosis or Compensated Cirrhosis Due to Nonalcoholic Steatohepatitis (NASH)
Acronym: ATLAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-454-4378
Record Dates: First submitted 2018-02-23; First posted 2018-02-28 (Actual); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — firsocostat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Selonsertib (SEL) (Experimental): Participants will receive SEL + placebo to match firsocostat 20 mg tablet + placebo to match cilofexor 30 mg tablet orally once daily for 48 weeks.
  Interventions: Drug: SEL; Drug: Placebo to match FIR; Drug: Placebo to match CILO
- Firsocostat (FIR) (Experimental): Participants will receive placebo to match SEL 18 mg tablet + FIR + placebo to match CILO 30 mg tablet orally once daily for 48 weeks.
  Interventions: Drug: FIR; Drug: Placebo to match CILO; Drug: Placebo to match SEL
- Cilofexor (CILO) (Experimental): Participants will receive placebo to match SEL 18 mg tablet + placebo to match FIR 20 mg tablet + CILO orally once daily for 48 weeks.
  Interventions: Drug: CILO; Drug: Placebo to match FIR; Drug: Placebo to match SEL
- Selonsertib (SEL) + Firsocostat (FIR) (Experimental): Participants will receive SEL + FIR + placebo to match CILO 30 mg tablet orally once daily for 48 weeks.
  Interventions: Drug: SEL; Drug: FIR; Drug: Placebo to match CILO
- Selonsertib (SEL) + Cilofexor (CILO) (Experimental): Participants will receive SEL + placebo to match FIR 20 mg tablet + CILO orally once daily for 48 weeks.
  Interventions: Drug: SEL; Drug: CILO; Drug: Placebo to match FIR
- Firsocostat (FIR) + Cilofexor (CILO) (Experimental): Participants will receive placebo to match SEL 18 mg tablet + FIR + CILO orally once daily for 48 weeks.
  Interventions: Drug: FIR; Drug: CILO; Drug: Placebo to match SEL
- Placebo (Experimental): Participants will receive placebo to match SEL 18 mg + placebo to match FIR 20 mg tablet + placebo to match CILO 30 mg tablet orally once daily for 48 weeks.
  Interventions: Drug: Placebo to match FIR; Drug: Placebo to match CILO; Drug: Placebo to match SEL

INTERVENTIONS:
Drug: SEL — 18 mg tablet administered orally once daily without regard to food
  Arms: Selonsertib (SEL); Selonsertib (SEL) + Cilofexor (CILO); Selonsertib (SEL) + Firsocostat (FIR)
Drug: FIR — 20 mg tablet administered orally once daily without regard to food
  Other Names: GS-0976
  Arms: Firsocostat (FIR); Firsocostat (FIR) + Cilofexor (CILO); Selonsertib (SEL) + Firsocostat (FIR)
Drug: CILO — 30 mg tablet administered orally once daily without regard to food
  Other Names: GS-9674
  Arms: Cilofexor (CILO); Firsocostat (FIR) + Cilofexor (CILO); Selonsertib (SEL) + Cilofexor (CILO)
Drug: Placebo to match FIR — Tablet administered orally once daily without regard to food
  Arms: Cilofexor (CILO); Placebo; Selonsertib (SEL); Selonsertib (SEL) + Cilofexor (CILO)
Drug: Placebo to match CILO — Tablet administered orally once daily without regard to food
  Arms: Firsocostat (FIR); Placebo; Selonsertib (SEL); Selonsertib (SEL) + Firsocostat (FIR)
Drug: Placebo to match SEL — Tablet administered orally once daily without regard to food
  Arms: Cilofexor (CILO); Firsocostat (FIR); Firsocostat (FIR) + Cilofexor (CILO); Placebo

SUMMARY:
The primary objectives of this study are:

* To assess the safety and tolerability of selonsertib (SEL), firsocostat (FIR) and cilofexor (CILO), administered alone or in combination, in participants with bridging fibrosis or compensated cirrhosis due to NASH
* To evaluate changes in liver fibrosis, without worsening of NASH

ELIGIBILITY:
Key Inclusion Criteria:

* Liver biopsy consistent with NASH and F3 or F4 in the opinion of the central reader
* In participants who have never had a liver biopsy, liver stiffness by FibroScan® ≥ 14.0 kPa and Enhanced Liver Fibrosis (ELF™) Test score ≥ 9.8 at Screening
* Screening laboratory parameters, as determined by the central laboratory:

  * Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min, as calculated by the Cockcroft-Gault equation
  * Hemoglobin A1c (HbA1c) ≤ 9.5%
  * Alanine aminotransferase (ALT) < 5 x Upper Limits of Normal (ULN)
  * Platelet count ≥ 125,000/μL

Key Exclusion Criteria:

* Prior history of decompensated liver disease including ascites, hepatic encephalopathy, or variceal bleeding
* Child-Pugh (CP) score > 6 at Screening, unless due to an alternative etiology such as Gilbert's syndrome or therapeutic anticoagulation
* Model for End-Stage Liver Disease (MELD) score > 12 at Screening, unless due to an alternate etiology such as therapeutic anticoagulation
* Other causes of liver disease based on medical history and/or centralized review of liver histology, including but not limited to: alcoholic liver disease, hepatitis B, hepatitis C, autoimmune disorders (eg, primary biliary cholangitis, primary sclerosing cholangitis, autoimmune hepatitis), drug-induced hepatotoxicity, Wilson disease, clinically significant iron overload, or alpha-1-antitrypsin deficiency requiring treatment
* History of liver transplantation
* Current or prior history of hepatocellular carcinoma

Note: Other protocol defined Inclusion/ Exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (101):
- United States (81):
  - The Institute for Liver Health, Chandler, Arizona
  - Mayo Clinic Arizona, Mayo Clinic Hospital, Phoenix, Arizona
  - Liver Wellness Center, Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - eStudySite, Chula Vista, California
  - Southern California Liver Center, Coronado, California
  - Fresno Clinical Research Center, Fresno, California
  - UCSD NAFLD Clinical Research Center, La Jolla, California
  - Ruane Clinical Research Group Inc., Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - California Liver Research Institute, Pasadena, California
  - Huntington Medical Research Institutes Liver Center, Pasadena, California
  - Inland Empire Liver Foundation, Rialto, California
  - University of California, Davis Medical Center (study visits), Sacramento, California
  - Medical Associates Research Group, San Diego, California
  - South Denver Gastroenterology, PC, Englewood, Colorado
  - Integrity Clinical Research, Doral, Florida
  - UF Hepatology Research at CTRB, Gainesville, Florida
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - IMIC Inc, Miami, Florida
  - Genoma Research Group, Miami, Florida
  - Florida Research Institute, Tampa, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Gastrointestinal Diseases Research, Columbus, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Northwestern University; Feinberg School of Medicine, Chicago, Illinois
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - Iowa Digestive Disease Center, P.C., Clive, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Delta Research Partners, LLC, Bastrop, Louisiana
  - Tulane University, New Orleans, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Digestive Disease Associates, PA, Catonsville, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health Systems, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Southern Therapy and Advanced Research (STAR) LLC, Ridgeland, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - Jubilee Clinical Research, Inc., Las Vegas, Nevada
  - Rutgers New Jersey Medical School- Doctors Office Center, Newark, New Jersey
  - Sandra Atlas Bass Center for Liver Diseases and Transplantation, Manhasset, New York
  - Icahn School of Medicine at Mount Sinai Beth Israel, New York, New York
  - Concorde Medical Group, PLLC, New York, New York
  - NYU Langone Health, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas Healthcare System Center for Liver Disease and Transplant, Charlotte, North Carolina
  - Duke University Medical Center, Duke South Clinics, Durham, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Consultants for Clinical Research wed, Cincinnati, Ohio
  - Hospital of the University of Pennsylvania- Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC - Center for Liver Diseases at the Thomas E. Starlz Institute, Pittsburgh, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Medical University of South Carolina (Liver Biopsy), Charleston, South Carolina
  - GHS Gastroenterology and Liver Center, Greenville, South Carolina
  - Gastro One, Germantown, Tennessee
  - Quality Medical Research, PLLC, Nashville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Pinnacle Clinical Research, PLLC, Austin, Texas
  - Austin Center for Clinical Research, Austin, Texas
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center Internal Medicine Digestive and Liver Diseases Clinical Trials, Dallas, Texas
  - Baylor College of Medicine - Advanced Liver Therapies, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Pinnacle Clinical Research, Live Oak, Texas
  - American Research Corporation at Texas Liver Institute, San Antonio, Texas
  - Intermountain Liver Disease and Transplant Center, Murray, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - California Pacific Medical Center - Sutter Pacific Medical Foundation San Francisco Center for Liver Disease Dept. of Transplant, Falls Church, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Bon Secours Richmond Community Hospital, Inc. d/b/a Bon Secours Liver Institute of Richmond, Richmond, Virginia
  - McGuire DVAMC, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Organ Transplant and Liver Center, Seattle, Washington
- Australia (12):
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Health, Monash Medical Centre, Clayton, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Melbourne Health, Royal Melbourne Hospital, Parkville, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
  - Royal Prince Alfred Hospital, Camperdown
  - St Vincent's Hospital Sydney, Darlinghurst
  - Austin Health, Heidelberg
  - The Alfred Hospital, Alfred Health, Melbourne
  - Westmead Hospital, Westmead
- Canada (5):
  - William Osler Health System-Brampton Civic Hospital, Brampton
  - University of Calgary Liver Unit (Heritage Medical Research Clinic), Calgary
  - Chronic Viral Illness Service McGill University Health Centre (MUHC)/ Royal Victoria Hospital, Montreal
  - Toronto General Hospital, Toronto
  - Toronto Liver Centre, Toronto
- Prince of Wales Hospital, Shatin, Hong Kong
- Auckland City Hospital, Auckland, New Zealand
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Loomba R, et al. Safety and efficacy of combination therapies including cilofexor/firsocostat in patients with bridging fibrosis and cirrhosis due to NASH: Results of the Phase 2b ATLAS trial [accepted for oral presentation]. European Association for the Study of the Liver (EASL); 2020; Virtual.
- [Result] Loomba R, Alkhouri N, Strasser S, Wong VWS, Schall RA, McColgan B, et al. Clinical utility and application of non-invasive tests of fibrosis in the selection of patients with advanced fibrosis due to NASH in the Phase 2 ATLAS trial (Poster SAT-315). EASL; 2019; Vienna, Austria.
- [Result] Loomba R, Alkhouri N, Patel K, Zhang J, McColgan BJ, Djedjos S, et al. Validation of Cutoffs for Controlled Attenuation Parameter with MRI-Proton Density Fat Fraction (PDFF) as a Reference Standard in Subjects with Nonalcoholic Steatohepatitis (NASH) Across Multiple Randomized, Controlled Trials (Poster 1727). American Association for the Study of Liver Diseases (AASLD); 2019; Boston, MA, USA.
- [Result] Loomba R, Alkhouri N, Noureddin M, Zhang J, McColgan BJ, Djedjos S, et al. Validation of the Diagnostic Accuracy of Magnetic Resonance Elastography (MRE) for the Detection of Advanced Fibrosis Due to Nash Across Multiple Phase 2 and 3 Clinical Trials (Poster 1728). AASLD; 2019; Boston, MA, USA.
- [Result] Alkhouri N, Strasser SI, Wong VWS, Aguilar R, Chuang J, Huss R, et al. Alcohol use is Underreported in Clinical Trials of NASH: Baseline Alcohol Biomarkers from a Phase 2 Clinical Trial (Poster 1765). AASLD; 2019; Boston, MA, USA.
- [Derived] Loomba R, Noureddin M, Kowdley KV, Kohli A, Sheikh A, Neff G, Bhandari BR, Gunn N, Caldwell SH, Goodman Z, Wapinski I, Resnick M, Beck AH, Ding D, Jia C, Chuang JC, Huss RS, Chung C, Subramanian GM, Myers RP, Patel K, Borg BB, Ghalib R, Kabler H, Poulos J, Younes Z, Elkhashab M, Hassanein T, Iyer R, Ruane P, Shiffman ML, Strasser S, Wong VW, Alkhouri N; for the ATLAS Investigators. Combination Therapies Including Cilofexor and Firsocostat for Bridging Fibrosis and Cirrhosis Attributable to NASH. Hepatology. 2021 Feb;73(2):625-643. doi: 10.1002/hep.31622. PMID 33169409

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States, Australia, Canada, Hong King and New Zealand. The first participant was screened on 21 Mar 2018. The last study visit occurred on 19 Nov 2019.
Pre-assignment Details: 950 participants were screened.
Groups:
- Selonsertib: Participants received selonsertib (SEL) 18 mg tablet + placebo to match firsocostat (FIR) 20 mg tablet + placebo to match cilofexor (CILO) 30 mg tablet orally once daily for 48 weeks.
- Firsocostat: Participants received placebo to match SEL 18 mg tablet + FIR 20 mg tablet + placebo to match CILO 30 mg tablet orally once daily for 48 weeks.
- Cilofexor: Participants received placebo to match SEL 18 mg + placebo to match FIR 20 mg tablet + CILO 30 mg tablet orally once daily for 48 weeks.
- SEL + FIR: Participants received SEL 18 mg tablet + FIR 20 mg tablet + placebo to match CILO 30 mg tablet orally once daily for 48 weeks.
- SEL + CILO: Participants received SEL 18 mg tablet + placebo to match FIR 20 mg tablet + CILO 30 mg tablet orally once daily for 48 weeks.
- FIR + CILO: Participants received placebo to match SEL 18 mg tablet + FIR 20 mg tablet + CILO 30 mg tablet orally once daily for 48 weeks.
- Placebo: Participants received placebo to match SEL 18 mg tablet + placebo to match FIR 20 mg tablet + placebo to match CILO 30 mg tablet orally once daily for 48 weeks.
Period: Overall Study
Arm/Group | Selonsertib | Firsocostat | Cilofexor | SEL + FIR | SEL + CILO | FIR + CILO | Placebo
Started | 39 | 40 | 41 | 80 | 78 | 78 | 39
Completed | 3 | 33 | 34 | 71 | 66 | 69 | 38
Not Completed | 36 | 7 | 7 | 9 | 12 | 9 | 1
Not completed — Randomized but Never Treated | 0 | 0 | 1 | 1 | 1 | 0 | 0
Not completed — Unknown Reason | 33 | 1 | 1 | 1 | 2 | 2 | 0
Not completed — Withdrew Consent | 1 | 3 | 1 | 4 | 4 | 4 | 1
Not completed — Adverse Event | 1 | 2 | 1 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1 | 3 | 0 | 0
Not completed — Investigator's Discretion | 0 | 1 | 1 | 2 | 0 | 0 | 0
Not completed — Non Compliance with Study Drug | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- Selonsertib: Participants received SEL 18 mg tablet + placebo to match FIR 20 mg tablet + placebo to match CILO 30 mg tablet orally once daily for 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Selonsertib | Firsocostat | Cilofexor | SEL + FIR | SEL + CILO | FIR + CILO | Placebo | Total
Number analyzed (Participants) | 39 | 40 | 40 | 79 | 77 | 78 | 39 | 392
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (10.4) | 60 (10.0) | 57 (10.2) | 59 (8.3) | 60 (9.0) | 61 (8.4) | 61 (8.2) | 60 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 29 | 49 | 51 | 48 | 27 | 253
  Male | 15 | 15 | 11 | 30 | 26 | 30 | 12 | 139
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of Race/ Ethnicity information.
  Participants
    Race: American Indian or Alaska Native | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 4
    Race: Asian | 7 | 3 | 0 | 3 | 4 | 5 | 3 | 25
    Race: Black | 0 | 1 | 0 | 1 | 2 | 2 | 1 | 7
    Race: Native Hawaiian or Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    Race: White | 30 | 35 | 40 | 73 | 68 | 68 | 35 | 349
    Race: Not Permitted | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Race: Other | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of Race/ Ethnicity information.
  Participants
    Ethinicity: Hispanic or Latino | 8 | 9 | 14 | 18 | 25 | 17 | 14 | 105
    Ethinicity: Not Hispanic or Latino | 31 | 31 | 26 | 60 | 52 | 60 | 25 | 285
    Ethinicity: Not Permitted | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  New Zealand | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Canada | 3 | 2 | 2 | 5 | 4 | 3 | 3 | 22
  Hong Kong | 2 | 0 | 0 | 3 | 2 | 2 | 1 | 10
  United States | 30 | 35 | 37 | 67 | 66 | 66 | 35 | 336
  Australia | 3 | 3 | 1 | 4 | 5 | 7 | 0 | 23
Diabetes Mellitus Status [Count of Participants; unit: Participants]
  Present | 26 | 30 | 27 | 57 | 58 | 57 | 27 | 282
  Absent | 13 | 10 | 13 | 22 | 19 | 21 | 12 | 110
Cirrhosis Status [Count of Participants; unit: Participants]
  Cirrhotic | 21 | 22 | 22 | 46 | 46 | 42 | 22 | 221
  Non-Cirrhotic | 18 | 18 | 18 | 33 | 31 | 36 | 17 | 171

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs)
Time Frame: First dose date up to 48 weeks plus 30 days
Population: The Safety Analysis Set included all participants who took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Selonsertib | Firsocostat | Cilofexor | SEL + FIR | SEL + CILO | FIR + CILO | Placebo
Number analyzed (Participants) | 39 | 40 | 40 | 79 | 77 | 78 | 39
percentage of participants | 84.6 | 85.0 | 92.5 | 88.6 | 96.1 | 91.0 | 79.5

2. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least one toxicity grade from baseline. Participants with any laboratory abnormality were reported.
Time Frame: First dose date up to 48 weeks plus 30 days
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Selonsertib | Firsocostat | Cilofexor | SEL + FIR | SEL + CILO | FIR + CILO | Placebo
Number analyzed (Participants) | 39 | 40 | 40 | 79 | 77 | 77 | 39
percentage of participants | 94.9 | 100.0 | 97.5 | 98.7 | 96.1 | 100.0 | 94.9

3. Primary Outcome: Percentage of Participants Who Achieved a ≥ 1-Stage Improvement in Fibrosis Without Worsening of NASH at Week 48
Description: Fibrosis improvement was defined as ≥ 1-stage decrease from baseline in fibrosis according to the NASH clinical research network classification (CRN) classification. Worsening of NASH was defined as ≥ 1-point increase from baseline in hepatocellular ballooning or lobular inflammation. The 95% CI was based on the Clopper-Pearson method.
Time Frame: Week 48
Population: Participants in the Full Analysis Set (included all participants who took at least 1 dose of study drug and were randomized into the study) with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Selonsertib | Firsocostat | Cilofexor | SEL + FIR | SEL + CILO | FIR + CILO | Placebo
Number analyzed (Participants) | 7 | 33 | 34 | 71 | 68 | 67 | 38
percentage of participants | 28.6 [3.7 to 71.0] | 12.1 [3.4 to 28.2] | 11.8 [3.3 to 27.5] | 15.5 [8.0 to 26.0] | 19.1 [10.6 to 30.5] | 20.9 [11.9 to 32.6] | 10.5 [2.9 to 24.8]
Statistical Analysis 1: Comparison: Firsocostat vs Placebo; Test type: Superiority; p = 0.9449, Mantel Haenszel — The p-value between each pair of treatment groups presented were obtained by the stratum-adjusted Mantel-Haenszel (MH) method, with baseline diabetes mellitus status and baseline cirrhosis status as stratification factors; Difference in percentages = 0.6, 95% CI 2-sided [-17.6 to 18.8] — The percentage difference and 95% C.I. presented were obtained by the stratum-adjusted MH method, with baseline diabetes mellitus status and baseline cirrhosis status as stratification factors
Statistical Analysis 2: Comparison: Cilofexor vs Placebo; Test type: Superiority; p = 0.9646, Mantel Haenszel — The p-value between each pair of treatment groups presented were obtained by the stratum-adjusted MH method, with baseline diabetes mellitus status and baseline cirrhosis status as stratification factors; Difference in percentages = 0.4, 95% CI 2-sided [-17.6 to 18.4] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: SEL + FIR vs Placebo; Test type: Superiority; p = 0.6219, Mantel Haenszel — [p-value comment as in outcome 3, analysis 2]; Difference in percentages = 3.7, 95% CI 2-sided [-10.9 to 18.3] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: SEL + CILO vs Placebo; Test type: Superiority; p = 0.2554, Mantel Haenszel — [p-value comment as in outcome 3, analysis 2]; Difference in percentages = 8.8, 95% CI 2-sided [-6.4 to 24.1] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: FIR + CILO vs Placebo; Test type: Superiority; p = 0.1658, Mantel Haenszel — [p-value comment as in outcome 3, analysis 2]; Difference in percentages = 10.8, 95% CI 2-sided [-4.5 to 26.1] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Firsocostat vs SEL + FIR; Test type: Superiority; p = 0.6963, Mantel Haenszel — [p-value comment as in outcome 3, analysis 2]; Difference in percentages = 3.2, 95% CI 2-sided [-12.9 to 19.4] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: Firsocostat vs FIR + CILO; Test type: Superiority; p = 0.2441, Mantel Haenszel — [p-value comment as in outcome 3, analysis 2]; Difference in percentages = 10.0, 95% CI 2-sided [-6.8 to 26.8] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: Cilofexor vs SEL + CILO; Test type: Superiority; p = 0.5229, Mantel Haenszel — [p-value comment as in outcome 3, analysis 2]; Difference in percentages = 5.2, 95% CI 2-sided [-10.7 to 21.0] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: Cilofexor vs FIR + CILO; Test type: Superiority; p = 0.2149, Mantel Haenszel — [p-value comment as in outcome 3, analysis 2]; Difference in percentages = 10.4, 95% CI 2-sided [-6.0 to 26.9] — [estimate comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: First dose date up to 48 weeks plus 30 days
Description: The Safety Analysis Set included all participants who took at least 1 dose of study drug.
Arm/Group | Selonsertib | Firsocostat | Cilofexor | SEL + FIR | SEL + CILO | FIR + CILO | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/40 | 0/40 | 0/79 | 1/77 | 0/78 | 0/39
Serious Adverse Events (participants affected / at risk) | 7/39 | 3/40 | 8/40 | 7/79 | 10/77 | 8/78 | 2/39
Other Adverse Events (participants affected / at risk) | 30/39 | 30/40 | 34/40 | 67/79 | 68/77 | 66/78 | 29/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selonsertib (N=39) | Firsocostat (N=40) | Cilofexor (N=40) | SEL + FIR (N=79) | SEL + CILO (N=77) | FIR + CILO (N=78) | Placebo (N=39)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 3 | 1 | 0 | 0 | 0
Colonic abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Incision site discharge (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Optic neuritis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression suicidal (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Selonsertib (N=39) | Firsocostat (N=40) | Cilofexor (N=40) | SEL + FIR (N=79) | SEL + CILO (N=77) | FIR + CILO (N=78) | Placebo (N=39)
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 1 | 5 | 0 | 2
Vision blurred (Eye disorders) | 0 | 1 | 0 | 1 | 4 | 6 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 1 | 4 | 1 | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 7 | 2 | 3 | 6 | 6 | 7 | 2
Abdominal pain lower (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3 | 1 | 6 | 7 | 5 | 5
Constipation (Gastrointestinal disorders) | 2 | 0 | 4 | 8 | 11 | 6 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 5 | 0 | 11 | 7 | 13 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 2 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 2 | 4 | 0
Nausea (Gastrointestinal disorders) | 3 | 6 | 3 | 20 | 10 | 10 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 10 | 2 | 2 | 1
Chest pain (General disorders) | 1 | 0 | 1 | 2 | 7 | 1 | 0
Fatigue (General disorders) | 5 | 7 | 3 | 14 | 9 | 8 | 3
Malaise (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 2 | 2 | 7 | 1 | 5 | 1
Pain (General disorders) | 0 | 2 | 0 | 0 | 1 | 2 | 1
Peripheral swelling (General disorders) | 3 | 0 | 0 | 2 | 1 | 3 | 0
Pyrexia (General disorders) | 0 | 3 | 1 | 5 | 2 | 3 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 2 | 2 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 8 | 7 | 2 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 5 | 4 | 0 | 2
Helicobacter infection (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 1 | 2
Influenza (Infections and infestations) | 0 | 3 | 0 | 1 | 4 | 5 | 1
Nasopharyngitis (Infections and infestations) | 2 | 4 | 6 | 3 | 3 | 9 | 5
Sinusitis (Infections and infestations) | 1 | 2 | 3 | 9 | 6 | 5 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 7 | 4 | 14 | 12 | 8 | 9
Urinary tract infection (Infections and infestations) | 6 | 3 | 5 | 9 | 9 | 6 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 2 | 1 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 2 | 1 | 3 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 3 | 9 | 4 | 6 | 5
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 2 | 2 | 1 | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4 | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3 | 2 | 8 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 5 | 9 | 7 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 3 | 4 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 4 | 4 | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4 | 7 | 4 | 7 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Carpal tunnel syndrome (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 5 | 2 | 4 | 8 | 9 | 3
Headache (Nervous system disorders) | 4 | 7 | 4 | 11 | 6 | 15 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2
Insomnia (Psychiatric disorders) | 1 | 1 | 2 | 1 | 5 | 2 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 2 | 1 | 2 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3 | 5 | 4 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 3 | 4 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 3 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 5 | 8 | 12 | 20 | 19 | 5
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 3 | 2 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 3 | 9 | 6 | 2 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 4 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/46/NCT03449446/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/46/NCT03449446/SAP_001.pdf